CLINICAL TRIAL: NCT01999283
Title: Effect of Group Pilates and Yoga Exercise Classes on Function, Range of Motion, Endurance, Postural Position, Medication Use and Balance in Adults With Chronic Cervical Pain
Brief Title: Effect of Group Pilates and Yoga Exercise Classes for Chronic Cervical Pain
Acronym: Pilates/Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Kim Dunleavy PhD, PT, OCS, Associate Professor Physical Therapy, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSUPT2013A
Record Dates: First submitted 2013-11-19; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Cervical Pain
Keywords: Cervical pain; yoga; pilates; exercise
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yoga Group Exercise (Active Comparator): Yoga group exercise will be taught by a licensed Physical Therapist. Groups consist of 4-8 individuals with 12 sessions once weekly over 12 weeks.
  Interventions: Other: Yoga Group Exercise
- Pilates Group Mat Exercise (Active Comparator): Pilates mat exercise will be taught by a licensed Physical Therapist with additional Rehabilitation Pilates certification.
  Interventions: Other: Pilates Group Mat Exercise
- Control (No Intervention): Wait Listed control group. Participants complete the same testing and were offered the option of attending the exercise classes on completion. The controls were not included in the exercise groups after completion.

INTERVENTIONS:
Other: Yoga Group Exercise — Yoga poses and postures modified to diminish stress on the cervical region and improve flexibility. Breathing and mind-body focus to address stress-related discomfort. A general Hatha yoga style will be used with components from Ashtanga Yoga. Intensity and range of motion will be progressively increased as tolerated.
  Arms: Yoga Group Exercise
Other: Pilates Group Mat Exercise — The Pilates mat exercises focus on both spinal muscle activation and stability, progressive endurance of the stabilizing muscles with arm and leg challenges and dynamic mobility. The exercises are progressed from more supported to anti-gravity position, slow increases in arm weights and flexibility.
  Arms: Pilates Group Mat Exercise

SUMMARY:
Exercise has been found to be effective in alleviating back and neck pain. Two exercise methods which are available in the community in a group format are Yoga and Pilates. While there is some research on the efficacy of these exercise methods for low back pain, there is no definitive research on the use of Yoga or Pilates group exercise for individuals with chronic cervical pain.This study investigated the effect of group Yoga and Pilates exercise compared to a wait-listed control group on impairments and function related to neck pain for individuals with chronic cervical pain.

DETAILED DESCRIPTION:
Individuals reporting chronic mild to moderate neck pain for more than 3 months were assigned to a pilates, yoga or wait-listed control group. The exercise group consisted of 12 one hour small group sessions instructed by experienced Physical Therapists with additional yoga or pilates training. Participants were evaluated at baseline, 6 weeks, and 12 weeks. Exercise participants also completed a follow up 6 weeks after completion.

ELIGIBILITY:
Inclusion Criteria:

* Able to attend at 12 exercise class sessions (once a week for an hour)
* Stable moderate to severe neck pain (3/10- 8/10) present for > 3 months
* Able to get up and down off the floor
* Able to ambulate in the community without an assistive device
* Medically stable and cleared to participate in exercise

Exclusion Criteria:

* Neck Pain that is easily aggravated with exercise
* Neurological symptoms in the arms or legs (numbness, tingling, weakness)
* History of recent whiplash, spine surgery, diagnosed osteoporosis, cervical stenosis with leg symptoms
* Any medical conditions which does not allow active exercise
* Unable to make medical decisions independently or have memory problems
* Regularly attending Pilates or Yoga classes or individual sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline Neck Disability Index | Baseline, 6 weeks, 12 weeks, 18 weeks
  Self reported Neck Disability Index questionnaire

SECONDARY OUTCOMES:
Change in Number of days of pain medication use in the past week | Baseline, week 6, week 12
  Self report
Change from baseline in Neck Pain Ratings (NPR) experienced on average over the past week | Baseline, week 6, week 12, week 18
  Average pain experienced over the past week (general, worst pain and experienced with functional activities - sustained positions, upper extremity movement, work, recreation)
Change from baseline Cervical range of motion measurements | Baseline, week 6, week 12, week 18
  Measured with the Cervical Range of Motion instrument (CROM)
Change from baseline differences between habitual and self corrected postural position | Baseline, week 6, week 12, week 18
  Sagittal plane position measured for Upper Cervical angle, forward head position, and thoracic width using the Cervical range of motion device.
Change from baseline in time for the Timed up and go test | Baseline, week 6, week 12, week 18
  Time to stand from a chair and walk to a standardized distance, return and sit down
Change from baseline Dynamic Gait Index score | Baselin, week 6, week 12, week 18
  Series of functional gait activities including walking, walking at different speeds, stepping over and around an obstacle, turning the head and tilting the head while walking scored by an observer.
Change from baseline in Activities Balance Confidence Scale score | Baseline, week 6, week 12, week 18
  Self reported confidence in maintaining balance for functional activities.

OTHER OUTCOMES:
Number of participants with identified potential for adverse drug responses | Baseline
  Descriptive analysis of number of participants with potential for adverse drug responses based on review of medication by Pharmacist
Identification of frequency of types of medication use in individuals with chronic neck pain | Baseline
  Descriptive analysis of medication used both for pain relief and co-morbidities
Frequency of types of potential adverse drug responses in patients with chronic mechanical neck pain | Baseline
  Identification of potential adverse drug responses by Pharmacist from medication review

CONTACTS AND LOCATIONS:
Overall Officials: Kim Dunleavy, PhD, PT, OCS, Principal Investigator — Wayne State University
Locations (4):
- United States (4):
  - Equilibrium Studio, Bloomfield Hills, Michigan
  - Wayne State University, Detroit, Michigan
  - Oakland Physical Therapy, Novi, Michigan
  - Older Persons Commission, Rochester, Michigan

REFERENCES:
- [Derived] Dunleavy K, Kava K, Goldberg A, Malek MH, Talley SA, Tutag-Lehr V, Hildreth J. Comparative effectiveness of Pilates and yoga group exercise interventions for chronic mechanical neck pain: quasi-randomised parallel controlled study. Physiotherapy. 2016 Sep;102(3):236-42. doi: 10.1016/j.physio.2015.06.002. Epub 2015 Aug 13. PMID 26435334